CLINICAL TRIAL: NCT04281797
Title: Intestinal Microbiome Composition Dynamics Over the Course of Kidney Transplantation, Liver Transplantation, Allogeneic Hematopoietic Stem Cells and Mesenchymal Stem Cells Transplantation
Brief Title: Intestinal Microbiome Dynamics in Solid Organ and Stem Cell Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology (Other Government)
Responsible Party: Principal Investigator, Ihar Iskrou, Head of Cell Transplants Division, Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology
Other Study IDs: Microbiome Minsk_1
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Transplantation Infection; Kidney Transplant; Complications; Stem Cell Transplant Complications; Liver Transplant; Complications; Microbial Colonization
Keywords: Microbiome; Gut microbiome; Stem cell transplantation; Kidney transplantation
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples. Microbial purified PCR-products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Kidney transplant recipients: Patients received kidney transplantation, with a baseline pre-transplant fecal sample and post-transplant samples collected. Standard transplantation procedures and precautions are being performed.
  Interventions: Diagnostic Test: Intestinal microbiome new generation sequencing
- HSCT-recipients: Patients received hematopoietic stem cells transplantation, with a baseline pre-transplant fecal sample and post-transplant samples collected. Standard transplantation procedures and precautions are being performed.
  Interventions: Diagnostic Test: Intestinal microbiome new generation sequencing
- MSCT-recipients: Patients received mesenchymal stem cells transplantation, with a baseline pre-transplant fecal sample and post-transplant samples collected. Standard transplantation procedures and precautions are being performed.
  Interventions: Diagnostic Test: Intestinal microbiome new generation sequencing
- Liver transplant recipients: Patients received liver transplantation, with a baseline pre-transplant fecal sample and post-transplant samples collected. Standard transplantation procedures and precautions are being performed.
  Interventions: Diagnostic Test: Intestinal microbiome new generation sequencing

INTERVENTIONS:
Diagnostic Test: Intestinal microbiome new generation sequencing — Fecal samples collected at baseline pre-transplant and post-transplant, new generation 16s RNA sequencing performed.

SUMMARY:
This is a pilot study designed to investigate the alterations in the gut microbiome that occur during the course of kidney transplantation, liver transplantation, allogeneic hematopoietic stem cells and mesenchymal stem cells transplantation in association with the clinical outcomes.

DETAILED DESCRIPTION:
This is a pilot study designed to investigate the dynamic changes in the intestinal microbiome that occur during the course of kidney transplantation, liver transplantation, allogeneic HSCs and mesenchymal stem cells transplantation. Four patient cohorts will be followed. Cohort A: patients receiving kidney transplantation. Cohort B: patients receiving hematopoietic stem cells transplantation. Cohort C: patients receiving mesenchymal stem cells transplantation. Cohort D: patients receiving liver transplantation. Included participants are defined as patients with at least three analyzable stool samples including a baseline sample before the transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled into kidney transplantation or HSCs transplantation or MSCs transplantation or liver transplantation programs with fecal samples collected over the course of their initial transplant hospitalization.
* Be willing and able to provide written informed consent for the study.

Exclusion Criteria:

* Patients were excluded from the study if their first sample was not collected prior to the start of transplantation procedure.
* Samples were excluded from the analysis if they were not aliquoted and stored frozen within 24 hours of collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment will include both patients with planned transplantations as well as recipients in urgent need of transplantation. The study coordinator may identify potential participants via direct referral from a treating physician, review of transplant lists and schedules.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | 1 month post-transplant
  Dynamics of gut microbiome composition over the course of transplantation (Shannon diversity index, Simpson index, abundance of main taxonomic phyla)

SECONDARY OUTCOMES:
Infectious complications after transplantation | 2 years post-transplant
  Incidence of infectious complications
Organ or tissue rejection | 2 years post-transplant
  Incidence of organ or tissue rejection

CONTACTS AND LOCATIONS:
Overall Officials: Igor Stoma, MD, PhD, Principal Investigator — Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology
Locations (1):
- Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoma I, Littmann ER, Peled JU, Giralt S, van den Brink MRM, Pamer EG, Taur Y. Compositional Flux Within the Intestinal Microbiota and Risk for Bloodstream Infection With Gram-negative Bacteria. Clin Infect Dis. 2021 Dec 6;73(11):e4627-e4635. doi: 10.1093/cid/ciaa068. PMID 31976518
- [Background] Stoma I, Karpov I, Iskrov I, Krivenko S, Uss A, Vlasenkova S, Lendina I, Cherniak V, Suvorov D. Decolonization of Intestinal Carriage of MDR/XDR Gram-Negative Bacteria with Oral Colistin in Patients with Hematological Malignancies: Results of a Randomized Controlled Trial. Mediterr J Hematol Infect Dis. 2018 May 1;10(1):e2018030. doi: 10.4084/MJHID.2018.030. eCollection 2018. PMID 29755707
- [Background] Stoma I, Karpov I, Krivenko S, Iskrov I, Milanovich N, Koritko A, Uss A. Mesenchymal stem cells transplantation in hematological patients with acute graft-versus-host disease: characteristics and risk factors for infectious complications. Ann Hematol. 2018 May;97(5):885-891. doi: 10.1007/s00277-018-3250-8. Epub 2018 Jan 29. PMID 29380038
- [Result] Igor Stoma, Mikhail Uss, Natalia Milanovich, Valentina Stoma, Tatiana Gubanova, Ekaterina Moduleva, Igor Iskrov & Anatoly Uss (2022) Biodiversity screening of gut microbiome during the allogeneic hematopoietic stem cell transplantation: data from the real-life clinical practice, All Life, 15:1, 547-554, DOI: 10.1080/26895293.2022.2074546